CLINICAL TRIAL: NCT01675440
Title: Medtronic CoreValve® U.S. Expanded Use Study
Brief Title: Safety & Efficacy Study of the Medtronic CoreValve® System-Treatment of Symptomatic Severe Aortic Stenosis With Significant Comorbidities in Extreme Risk Subjects Who Need Aortic Valve Replacement
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 10050361DOC
Record Dates: First submitted 2012-08-22; First posted 2012-08-30 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Severe (≥3-4+) Mitral Valve Regurgitation: Mitral valve regurgitation ≥3-4+
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Severe (≥3-4+) Tricuspid Valve Regurgitation: Tricuspid valve regurgitation ≥3-4+
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- End Stage Renal Disease (ESRD): End stage renal disease requiring renal replacement therapy or a creatinine clearance (CRCL) <20 cc/min, but not on dialysis
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Low Gradient Low Output Aortic Stenosis: Low gradient low output aortic stenosis
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Failed Bioprosthetic Surgical Aortic Valve: Stenosed, insufficient or combined bioprosthetic surgical aortic valve failure
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- 2 or More Conditions: 2 or more of the listed conditions
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)

SUMMARY:
To evaluate the safety and efficacy of the Medtronic CoreValve® System for the treatment of symptomatic severe aortic stenosis in subjects with significant comorbidities in whom the risk of surgical aortic valve replacement has a predicted operative mortality or serious, irreversible morbidity risk of ≥50% at 30 days.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and effectiveness of the Medtronic CoreValve® System (MCS) in a subset of subjects excluded from the U.S. Extreme Risk Pivotal Trial population due to one or more additional co-morbidities, as measured by a composite of all-cause death or major stroke at 12 months, in the treatment of symptomatic severe aortic stenosis in subjects necessitating aortic valve replacement. Subjects enrolled in this study have a predicted operative mortality or serious, irreversible morbidity risk of ≥50% at 30 days associated with surgical aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have co-morbidities such that one cardiologist and two cardiac surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement. Specifically, the predicted operative risk of death or serious, irreversible morbidity is ≥ 50% at 30 days.
* Subjects must meet all of the criteria under at least one of the sub-groups 2a-c:

  a. Senile degenerative aortic valve stenosis and i. At least one of the following co-morbid conditions:
  1. Severe (≥3-4+) mitral valve regurgitation as measured by echocardiography
  2. Severe (≥3-4+) tricuspid valve regurgitation as measured by echocardiography
  3. End-stage renal disease requiring renal replacement therapy (Stage 5 of the KDOQI CKD Classification) or creatinine clearance <20cc/min but not requiring renal replacement therapy

     AND

     ii. mean gradient > 40 mmHg or jet velocity greater than 4.0 m/sec by either resting or dobutamine stress echocardiogram (if the LVEF < 50%), or simultaneous pressure recordings at cardiac catheterization either resting or with dobutamine stress (if the LVEF < 50%) AND iii. an initial aortic valve area of ≤ 0.8 cm2 (or aortic valve area index ≤0.5 cm2/m2) by resting echocardiogram or simultaneous pressure recordings at cardiac catheterization

     AND/OR

     b. Low gradient, low output aortic stenosis as defined by the presence of all three of the following i. In the presence of LVEF <50%, absence of contractile reserve, a mean gradient ≥25mmHg and <40mmHg AND jet velocity less than 4.0m/sec with dobutamine stress echocardiography or simultaneous pressure recordings at cardiac catheterization OR In the presence of LVEF ≥50%, a mean gradient ≥25mmHg and <40mmHg AND jet velocity less than 4.0 m/sec, by echocardiography or simultaneous pressure recordings at cardiac catheterization AND ii. an initial aortic valve area of ≤0.8 cm2 (or aortic valve area index ≤0.5 cm2/m2) by resting echocardiogram or simultaneous pressure recordings at cardiac catheterization AND iii. radiographic evidence of severe aortic valve calcification AND/OR c. Failed bioprosthetic surgical aortic valve
* Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater.
* The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the IRB of the respective clinical site.
* The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

Clinical

* Evidence of an acute myocardial infarction ≤30 days before the MCS TAVI procedure.
* Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the MCS TAVI procedure
* Blood dyscrasias as defined: leukopenia (WBC <1000mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy.
* Untreated clinically significant coronary artery disease requiring revascularization.
* Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
* Need for emergency surgery for any reason.
* Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% as measured by resting echocardiogram.
* Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
* Active Gastrointestinal (GI) bleeding that would preclude anticoagulation.
* A known hypersensitivity or contraindication to all anticoagulation/antiplatelet regimens (including ability to be anticoagulated for the index procedure), nitinol, or [allergic] sensitivity to contrast media which cannot be adequately pre-medicated.
* Ongoing sepsis, including active endocarditis.
* Subject refuses a blood transfusion.
* Life expectancy <12 months due to associated non-cardiac co-morbid conditions.
* Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
* Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
* Currently participating in an investigational drug or another device study.
* Symptomatic carotid or vertebral artery disease.

Anatomical

Subject has a:

* Native aortic annulus size <18 mm or >29 mm per the baseline diagnostic imaging (not applicable for TAV in SAV subjects) OR
* Surgical bioprosthetic annulus <17mm or >29mm i. Stented SAV per the manufactured labeled inner diameter OR ii. Stentless SAV per the baseline diagnostic imaging
* Subject has a pre-existing prosthetic heart valve with a rigid support structure in either the mitral or pulmonic position:

  1. that could affect the implantation or function of the study valve OR
  2. the implantation of the study valve could affect the function of the pre-existing prosthetic heart valve
* Moderate to severe mitral stenosis.
* Mixed aortic valve disease: aortic stenosis and aortic regurgitation with predominant aortic regurgitation, (AR is moderate-severe to severe (≥3-4+))(except for failed surgical bioprothesis)
* Hypertrophic obstructive cardiomyopathy.
* Echocardiographic evidence of new or untreated intracardiac mass, thrombus or vegetation.
* Severe basal septal hypertrophy with an outflow gradient.
* Aortic root angulation (angle between plane of aortic valve annulus and horizontal plane/vertebrae) >70° (for femoral and left subclavian/axillary access) and >30° (for right subclavian/axillary access).
* Ascending aorta that exceeds the maximum diameter for any given native or surgical bioprosthetic* aortic annulus size (see table below) Aortic Annulus Diameter/ Ascending Aorta Diameter, 18 mm* - 20 mm/ >34 mm, 20 mm - 23 mm/ >40 mm, 23 mm - 27 mm/ >43 mm, 27 mm - 29 mm/ >43 mm,

  * 17mm for surgical bioprosthetic aortic annulus
* Congenital bicuspid or unicuspid valve verified by echocardiography (Not applicable for TAV in SAV subjects).
* Sinus of valsalva anatomy that would prevent adequate coronary perfusion.
* Degenerated surgical bioprothesis presents with a significant concomitant perivalvular leak (between prothesis and native annulus), is not securely fixed in the native annulus, or is not structurally intact (e.g. wireform frame fracture) (ONLY FOR TAV in SAV subjects)
* Degenerated surgical bioprothesis presents with a partially detached leaflet that in the aortic position may obstruct a coronary ostium (ONLY FOR TAV in SAV subjects)

Vascular

* Transarterial access not able to accommodate an 18Fr sheath.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with symptomatic severe aortic stenosis requiring aortic valve replacement, with predicted operative mortality or serious, irreversible morbidity risk of ≥ 50% at 30 days, and at least one of the following conditions:
  * Severe (≥3-4+) mitral valve regurgitation
  * Severe (≥3-4+) tricuspid valve regurgitation
  * End stage renal disease (ESRD) requiring renal replacement therapy or creatinine clearance <20cc/min, but not requiring renal replacement therapy
  * Low gradient, low output aortic stenosis
  * Failed bioprosthetic surgical aortic valve
  * 2 or more conditions (listed above)
Sampling Method: Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2012-08; Primary Completion 2016-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
All-cause Mortality or Major stroke | 12 months
  All-cause Mortality or Major Stroke

SECONDARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Event (MACCE) Event Rate | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  MACCE is defined as a composite of: • All-Cause Death • Myocardial Infarction (MI) • All Stroke • Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
The Occurrence of individual MACCE Components | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  Individual MACCE Components Include: - All Cause Mortality - MI - All stroke - Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Major Adverse Events (MAEs) | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  MAEs Include: •MACCE •Acute Kidney Injury •Cardiac Tamponade •Prosthetic Valve Dysfunction •Cardiogenic Shock •Valve Endocarditis •Life-Threatening, Disabling or Major Bleeding •Major Vascular Complication •Cardiac Perforation •Device Migration/Valve Embolism
Conduction Disturbance Requiring Permanent Pacemaker Implantation | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  The incidence of conduction disturbance requiring permanent pacemaker implantation
Change in NYHA Class | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  Change from baseline (continuous variable). A positive number corresponds to NYHA worsening; a negative number corresponds to NYHA improvement.
Change in Distance Walked During 6-minute Walk Test (6MWT) from Baseline | 30 days and 12 months
  Change in distance walked during 6MWT from baseline
Ratio of Days Alive Out of Hospital Versus Total Days Alive | 12 months
Quality of Life (QoL) Change from Baseline | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  QoL change from baseline using the following measures: •Kansas City Cardiomyopathy Questionnaire (KCCQ) •SF-12 •EuroQoL
Echocardiographic Assessment of Valve Performance | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  Using the following measures: • Transvalvular mean gradient • Effective orifice area (EOA) •degree of aortic valve regurgitation
Aortic Valve Disease Hospitalization | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  The number of subjects re-hospitalized after the initial procedure
Cardiovascular Deaths and Valve-related Deaths | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  The number of cardiovascular deaths and valve-related deaths
Strokes | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  The number of subjects with strokes and TIAs
Index Procedure Related Major Adverse Events (MAEs) | Procedure
  Index procedure-related MAE events will be summarized
Length of Index Procedure Hospital Stay | Number of days from admission to discharge
  The length of index procedure hospital stay will be summarized
Device Success | Number of days from admission to discharge
  Defined as: 1) Successful vascular access, delivery and deployment of the device, and successful retrieval of the delivery system, 2) Correct position of the device in the proper anatomical location (placement in the annulus with no impedance on device function), 3) Intended performance of the prosthetic valve (aortic valve area > 1.2 cm2 for 26, 29 and 31mm valves, ≥ 0.9 cm2 for 23mm valve (by echocardiography using the continuity equation) and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/sec, without moderate or severe prosthetic valve aortic regurgitation) 4) Only one valve implanted in the proper anatomical location. For TAV in SAV subjects, only # 1, 2 and 4 will be used to calculate device success.
Procedural Success | Number of days from admission to discharge
  Defined as device success and absence of in-hospital MACCE
Evidence of Prosthetic Valve Dysfunction | 30 days, 6 months, 12 months and annually thereafter up to 5 years
  PVD was defined according to VARC using the site reported echocardiography assessments including aortic regurgitation (AR) and aortic stenosis (AS) evaluations. Total AR reported as moderate or severe was considered PVD. AS was defined as significant stenosis and considered PVD if one of the following was met: •Peak velocity > 4 m/s •Mean gradient > 35 mmHg •EOA < 0.8 cm2 •TVIV1 / TVIV2 < 0.25

CONTACTS AND LOCATIONS:
Overall Officials: David H Adams, Principal Investigator — Mount Sinai Health System
Locations (43):
- United States (43):
  - Banner Good Samaritan, Phoenix, Arizona
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - University of Southern California University Hospital, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center / Georgetown Hospital, Washington D.C., District of Columbia
  - University of Miami Health System / Jackson Memorial Hospital, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Cardiovascular Institute of the South/Terrebonne General, Houma, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Detroit Medical Center Cardiovascular Institute, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Morristown Memorial Hospital, Morristown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University - Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals - Case Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center - The Richard M. Ross Heart Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital - The Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - St. Luke's Medical Center - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Butala NM, Song Y, Shen C, Cohen DJ, Yeh RW. Effect of intensive versus limited monitoring on clinical trial conduct and outcomes: A randomized trial. Am Heart J. 2022 Jan;243:77-86. doi: 10.1016/j.ahj.2021.09.002. Epub 2021 Sep 14. PMID 34529944
- [Derived] Dauerman HL, Deeb GM, O'Hair DP, Waksman R, Yakubov SJ, Kleiman NS, Chetcuti SJ, Hermiller JB Jr, Bajwa T, Khabbaz K, de Marchena E, Salerno T, Dries-Devlin JL, Li S, Popma JJ, Reardon MJ. Durability and Clinical Outcomes of Transcatheter Aortic Valve Replacement for Failed Surgical Bioprostheses. Circ Cardiovasc Interv. 2019 Oct;12(10):e008155. doi: 10.1161/CIRCINTERVENTIONS.119.008155. Epub 2019 Oct 14. PMID 31607151